CLINICAL TRIAL: NCT02701478
Title: Assessment of the Intraoperative Analgesic Effect of 50%/50% N2O/O2 Inhalation by the Pain Index ANI Following a Standardized Electrical Stimulus in Patients Under Anesthesia. Comparison to the New NoL Analgesic Index.
Brief Title: ANI and NoL Index Variations After Standard Nociceptive Stimulus at 0, 50, 25 % of Inhaled N2O in the Anesthetic Mixture
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Maisonneuve-Rosemont Hospital (Other)
Responsible Party: Principal Investigator, Philippe Richebé, Full Professor of Anesthesiology and Pain medicine, Maisonneuve-Rosemont Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 15064
Record Dates: First submitted 2016-03-02; First posted 2016-03-08 (Estimated); Last update posted 2016-11-18 (Estimated); Status verified 2016-11

CONDITIONS: Pain
MeSH Terms: conditions — Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- N2O exposure (Other): There is only one arm in this study. All patients under General Anesthesia are exposed to 4 different doses or concentrations of inhaled N2O that is combined with the anesthetic desflurane. Each patient will be submitted to the standard nociceptive stimulus when inhaled N2O is at 0, 50, 25, and finally back to 0%. ANI and NoL Indices variations between "before stimulus" and "after stimulus" at each N2O concentration will be assessed and compared. This will allow to demonstrate an analgesic effect (less variations of ANI and NoL) when inhaled N2O is high (50%) testifying for the analgesic effect of this gas N2O.
  Interventions: Drug: N2O exposure

INTERVENTIONS:
Drug: N2O exposure — The aim of this study is to evaluate the nociceptive response to a standardized forearm electrical stimulus applied to patients under GA, during surgery, at different End-Tidal concentrations of N2O (ET-N2O: 0%-50%-25%-0%), and to see if ANI and NoL indices show less pain when inhaled N2O is higher.
  Other Names: N2O

SUMMARY:
N2O has been used during general anesthesia (GA) for more than 100 years. It is known to have anesthetic agents sparing effect. But small is know on his real analgesic effect during GA. So far, the only way to monitor pain during GA was based on vital signs that are not specific and not sensitive. Few devices tried to evaluated pain under GA during the last 2 decades. More recently, better devices were proposed such as the Physiodoloris device and the PMD200 device. The first offers an index called ANI based on heart rate variability (HRV) assessment. The second offers the NoL index based on the analysis of 5 parameters. The aim of the present study is to evaluate quantitatively the analgesic index of N2O during GA using the two indices ANI and NoL.

DETAILED DESCRIPTION:
Title: Assessment of the intraoperative analgesic effect of 50%/50% Nitrous Oxide / Oxygen inhalation by the pain index ANI following a standardized electrical forearm stimulus in patients undergoing laparotomies under general anesthesia and with an intraoperative active epidural analgesia. Comparison to the new NoL analgesic index.

Objectives: To observe the variations of the intraoperative pain indexes ANI and NoL after a classical and standardized electrical stimulation of the forearm (applied with the commonly used nerve stimulator we use for muscle relaxation monitoring) at different concentrations of inhaled Nitrous Oxide (N2O) (from 0% to 50%, concentrations that are commonly used in daily anesthesia). This will allow a quantification of the analgesic effect of N2O.

Study Design: Prospective, open label, observational and descriptive study Subject Population: Adult patients scheduled to undergo abdominal surgery by laparotomy under general anesthesia with an active intraoperative epidural analgesia Sample Size: 40 patients will be evaluated in this study Study Duration: 1 year Study Center: Maisonneuve-Rosemont Hospital, Montreal, Quebec, Canada Adverse Events: None expected

ELIGIBILITY:
Inclusion Criteria:

* ASA status I, II or III
* Patients aged 18 to 70 years
* Laparotomy for gynecological or bowel surgery
* Duration and type of surgery requiring an epidural analgesia via an epidural catheter placed prior the general anesthesia induction and an arterial line placed after induction of general anesthesia

Exclusion Criteria:

* When 100% O2 ventilation is required during anesthesia (except for the induction phase during which all the patients receive O2 100%).
* Patients having received intraocular injection of gas (such as SF6, C3F8, C2F6) within 3 months prior to the present surgery.
* Any condition where internal entrapped air could expand and become dangerous, such as:

  * head injury within 6 months prior to surgery
  * maxillofacial injuries within 6 months prior to surgery
  * pneumothorax within 6 months prior to surgery
  * gas embolism within 6 months prior to surgery
  * decompression sickness within 6 months prior to surgery
  * bubbles of emphysema known for this patient
  * middle ear, inner ear and sinus surgery
  * major abdominal distension/occlusion and emergent surgery for intestinal obstruction
  * if air has been injected into the epidural space to determine the placement of the needle for epidural anesthesia (only saline is used in our center for the loss of resistance technique to place the catheter into the epidural space)

Any contra-indication or patient's refusal for epidural placement

* Unexpected difficult airway requesting excessive, possibly painful airway manipulations.
* Unexpected surgical complications requiring strong haemodynamic support (transfusions, volume challenges, vasopressors, inotropic drugs).

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2016-01; Primary Completion 2016-12 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
ANI variation after stimulation in patients under GA at End-Tidal N2O 0% and 50%. | First stimulus is applied when the patient breaths 0% N2O in his anesthesia mixture. Second stimulus is applied at 50% End-Tidal N2O in the anesthesia mixture during the surgery.
  The same patient is anesthetized without N2O in the gas mixture first. The first standard stimulus is applied on the forearm of the patient when the N2O concentration in the anesthesia mixture is at 0%. ANI response to the stimulus is recorded. Then N2O is slowly increased to reached et-N2O 50% in the anesthesia mixture. Then, at ET-N2O 50%, the same standard stimulus is applied and ANI variations registered.

SECONDARY OUTCOMES:
NoL index variation after electrical stimulation in patients under GA atEnd-Tidal N2O 0% and 50%. | First stimulus is applied when the patient breaths 0% N2O in his anesthesia mixture. Second stimulus is applied at 50% End-Tidal N2O in the anesthesia mixture during the surgery.
  The same patient is anesthetized without N2O in the gas mixture first. The first standard stimulus is applied on the forearm of the patient when the N2O concentration in the anesthesia mixture is at 0%. NoL response to the stimulus is recorded. Then N2O is slowly increased to reached et-N2O 50% in the anesthesia mixture. Then, at ET-N2O 50%, the same standard stimulus is applied and NoL variations registered.
ANI and NoL indices variations after the same standard stimulus when ET-N2O is slowly decreased from 50% to 25%, , then to 0%. | Within the same anesthesia and surgery
  During the surgery, for primary and secondary objectives, N2O will be at 0, then 50%.
  For these secondary objectives, N2O inhaled concentration in teh anesthetic mixture will be set at 25% and then again at 0% and the same standard stimulus will be applied and ANI and NoL responses recorded and compared to the ones gotten at 50% .

CONTACTS AND LOCATIONS:
Overall Officials: Philippe Richebe, MD PhD, Principal Investigator — Maisonneuve-Rosemont Hospital
Locations (1):
- Hopital Maisonneuve Rosemont, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Coulombe MA, Decary E, Maximos S, Brulotte V, Drolet P, Tanoubi I, Issa R, Zaphiratos V, Verdonck O, Fortier LP, Godin N, Idrissi M, Raft J, Richebe P. Assessing the antinociceptive effect of nitrous oxide to tetanic stimulation in anaesthetised patients with new intra-operative nociception monitors: An observational study. Eur J Anaesthesiol. 2021 May 1;38(5):512-523. doi: 10.1097/EJA.0000000000001431. PMID 33399383